CLINICAL TRIAL: NCT06989034
Title: Sensory Processing Abilities in Relation to Postural Stability and Selective Motor Control in Children With Hemiplegia.
Brief Title: Sensory Processing, Postural Stability, and Selective Motor Control in Children With Hemiplegia
Acronym: HeSPoM
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Fathi Fouad Hussein, Teaching Assistant, Cairo University
Other Study IDs: P.T.REC/012/004244
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy, Hemiplegic; Sensory Processing Disorder; Postural Balance; Motor Skills Disorders
Keywords: sensory processing abilities; Postural stability; selective voluntary motor control; unilateral cerebral palsy; child sensory profile 2
MeSH Terms: conditions — Cerebral Palsy; Motor Skills Disorders | interventions — Sp2 Transcription Factor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The hemiplegic cerebral palsy (CP) group: The hemiplegic cerebral palsy (CP) group consists of 30 children diagnosed with spastic hemiplegic CP, a type of CP characterized by motor impairment predominantly on one side of the body. These children were aged between 6 and 10 years and had GMFCS levels I or II, indicating mild to moderate functional limitations. They exhibited mild spasticity, as indicated by Modified Ashworth Scale scores of 1 or 1+, and were able to follow simple instructions. The hemiplegic CP group was included to investigate sensory processing, postural stability, and selective voluntary motor control (SVMC) impairments associated with spastic hemiplegia.
  Interventions: Other: Child Sensory Profile 2 (SP2) for Sensory processing abilities; Other: HUMAC Balance System for Postural stability evaluation; Other: Selective Motor Control Evaluation for the upper and lower extremities
- typically developing children (TDC) group: The control group consisted of 30 typically developing children (TDC) who were matched to the hemiplegic CP group based on age and sex. The control group served as a comparison to the CP group, allowing for the evaluation of typical sensory processing, postural stability, and selective voluntary motor control patterns in children without any clinical motor impairments. The children in the control group were expected to perform within typical developmental ranges for sensory and motor function, providing a baseline for assessing the motor and sensory processing deficits in the hemiplegic CP group.
  Interventions: Other: Child Sensory Profile 2 (SP2) for Sensory processing abilities; Other: HUMAC Balance System for Postural stability evaluation; Other: Selective Motor Control Evaluation for the upper and lower extremities

INTERVENTIONS:
Other: Child Sensory Profile 2 (SP2) for Sensory processing abilities — Sensory processing abilities are evaluated using the Child Sensory Profile 2 (SP2), an 86-item caregiver questionnaire assessing six sensory systems (auditory, visual, touch, movement, body position, and oral) and three behavioral domains (conduct, social-emotional, and attentional).
Other: HUMAC Balance System for Postural stability evaluation — Postural stability is assessed using the HUMAC Balance System, incorporating tests such as:
  * The Modified Clinical Test of Sensory Integration of Balance (mCTSIB)
  * Limits of Stability (LOS) at difficulty levels 4 and 6
  * Center of Pressure (COP) metrics
Other: Selective Motor Control Evaluation for the upper and lower extremities — Selective voluntary motor control is evaluated using the following tools:
  * Test of Arm Selective Control (TASC) for the upper extremities
  * Selective Control Assessment of the Lower Extremity (SCALE) for the lower extremities

SUMMARY:
The goal of this observational case-control study is to examine the relationship between sensory processing abilities, postural stability, and selective motor control (SMC) in children aged 6-10 years with hemiplegic cerebral palsy (CP). The study compares outcomes in children with hemiplegic CP to age-matched typically developing children (TDC). It aims to determine how differences in sensory processing may relate to motor control and balance deficits in this population.

DETAILED DESCRIPTION:
This study investigated the associations between sensory processing abilities, postural stability, and selective voluntary motor control (SVMC) in children diagnosed with hemiplegic cerebral palsy (CP), and compared these findings to age-matched typically developing children (TDC). Thirty children with hemiplegic CP and thirty TDC aged 6-10 years were recruited based on predefined inclusion and exclusion criteria. Children with CP were selected from the outpatient clinic at the Faculty of Physical Therapy, Cairo University.

The study used validated clinical tools: the Child Sensory Profile 2 (SP2) to assess sensory processing abilities across multiple sensory systems and behavioral domains; the HUMAC balance system to evaluate postural stability through modified clinical tests of sensory integration, center of pressure testing, and limits of stability assessments; the Test of Arm Selective Control (TASC) and the Selective Control Assessment of the Lower Extremity (SCALE) to evaluate upper and lower limb SVMC, respectively.

All participants were assessed in a controlled clinical setting, and statistical comparisons were made between the two groups. The study also examined the correlations between sensory profile data and motor/postural outcomes. Ethical approval was obtained, and informed consent was secured from all caregivers. The results are intended to provide insights into the interaction between sensory processing and motor control deficits in children with hemiplegia and to support clinicians in tailoring interventions based on sensory-motor integration profiles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spastic hemiplegic cerebral palsy
* Age between 6 and 10 years
* GMFCS levels I or II
* Modified Ashworth Scale score of 1 or 1+ (mild spasticity)
* Ability to follow simple instructions
* Caregiver with sufficient English language proficiency

Exclusion Criteria:

* Botulinum toxin injections within the past 6 months
* Visual or auditory impairments
* Orthopedic or neurosurgical intervention to limbs or spine
* Musculoskeletal deformities
* History of seizures

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population divided into two groups. The first group includes 30 children diagnosed with spastic hemiplegic cerebral palsy (CP), a condition characterized by motor impairments affecting one side of the body due to early brain damage. These children are recruited from the outpatient clinic of the Faculty of Physical Therapy, Cairo University.
  The second group includes 30 age- and sex-matched typically developing children (TDC) who have no known neurological, orthopedic, or sensory processing disorders. These children are selected from mainstream schools in Luxor Governorate and are expected to exhibit typical development in sensory processing, motor control, and postural stability.
  The children in the CP group are part of a clinical setting with prior diagnoses and care, while the TDC group is sourced from an educational setting. The study aims to compare sensory processing abilities, postural stability, and selective motor control
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
ensory Profile 2 (SP2) Total and Subscale Scores | Single assessment session (within a 1-day visit)
  Scores across sensory domains and behavioral responses will be compared between groups and correlated with motor outcomes.
HUMAC Balance Scores (COP, LOS, mCTSIB) | Single assessment session (within a 1-day visit)
  Quantitative balance parameters will be analyzed between groups.
TASC and SCALE Scores | Single assessment session (within a 1-day visit)
  Selective motor control scores (range 0-2 per joint movement) will be summed and analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- outpatient clinic, Faculty of Physical Therapy, Cairo University, Giza, Cairo Governorate, Egypt